CLINICAL TRIAL: NCT04065243
Title: Metabolic Changes in Response to Experimental Overfeeding: A Randomized Intervention Study
Brief Title: Experimental Overfeeding in Humans
Acronym: ExpO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Christoffer Clemmensen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ExpO
Record Dates: First submitted 2019-08-08; First posted 2019-08-22 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Overfed; Obesity
MeSH Terms: conditions — Overnutrition; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Body weight and other anthropometric data are not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Subjects in this group will have a daily energy intake equivalent of 100 % of their calculated normal daily energy intake.
  Interventions: Other: Isocaloric diet
- Overfed group (Experimental): Subjects in this group will have a daily energy intake equivalent of 150 % of their calculated normal daily energy intake.
  Interventions: Other: Overfeeding diet

INTERVENTIONS:
Other: Overfeeding diet — Two weeks of overfeeding
  Arms: Overfed group
Other: Isocaloric diet — Two weeks of isocaloric weight maintenance
  Arms: Control group

SUMMARY:
The objective of this study is to determine the homeostatic mechanisms that counteract weight gain in response to experimental overfeeding.

DETAILED DESCRIPTION:
The homeostatic regulation of body weight implies that biological processes have evolved to protect energy stores from changes to the food environment. Accordingly, many individuals remain remarkably weight stable over years without carefully considering how much they eat or how much energy they expend, which has given rise to the theory that body weight is regulated around an individual biological 'set point'. Notably, overfeeding humans in experimentally controlled conditions, support this phenomenon, but the underlying mechanisms are unknown.

To systematically map out the components of the overfed state, the investigators will execute a 2-week randomized controlled overfeeding trial in lean and overweight individuals. The trial is preceded by a 1-week lead-in period and followed by a 2-wk controlled ad libitum study period. The comparison between lean and overweight subjects, men and women, enables the determination of whether a differential response in overfeeding-induced signals is present in relation to BMI and sex.

ELIGIBILITY:
Inclusion Criteria:

* Male or female otherwise healthy subjects
* 20-40 years of age
* BMI (Body mass index) between 22-30 kg/m2

Exclusion Criteria:

* Present or previous cardiovascular disease, diabetes or thyroid-disease
* smoking
* more than 3 hours of planned physical activity per week

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in blood protein patterns using proteomics 1 week before, during 2 weeks of overfeeding and 2 weeks after overfeeding | 5 weeks
  Blood will be collected for proteomics at screening, at baseline, during the overfeeding intervention and during the 2-week ad libitum intervention. Samples will be measured using LCMS instrumentation consisting of a nanoelectrospray ion source to a Q Exactive HF mass spectrometer.
Changes in blood peptide patterns using peptidomics 1 week before, during 2 weeks of overfeeding and 2 weeks after overfeeding | 5 weeks
  Blood will be collected for peptidomics at screening, at baseline, during the overfeeding intervention and during the 2-week ad libitum intervention. Samples will be measured using LCMS instrumentation consisting of a nanoelectrospray ion source to a Q Exactive HF mass spectrometer.

SECONDARY OUTCOMES:
Body weight | 5 weeks
  Body weight will be measured (in kilograms) daily during the intervention using electronic Fitbit Aria 2 weight scale.
Fat biopsy from subcutaneous adipose tissue before and after 2 weeks of overfeeding | 2 weeks
  Fat biopsies are obtained using Bergström biopsy needle from subcutaneous adipose tissue in the abdominal region before and after 14 days of overfeeding to assess regulated enzymes and proteins.
Microdialysate from subcutaneous adipose tissue before and after 2 weeks of overfeeding. The samples will be used for detection of known and unknown secreted factors | 2 weeks
  Microdialysates are collected from micro dialysis catheters inserted into the subcutaneous adipose tissue in the abdominal region before and after 14 days of overfeeding to assess regulated enzymes and proteins.
Body composition in 40 subjects before and after overfeeding | 3 weeks
  Body composition will be measured using Dual-Energy X-ray Absorptiometry (DXA) at screening (1 week before baseline), at baseline and after 14 days of overfeeding. The DXA scan enables the detection of body lean mass and body fat mass in kg.
Mixed meal test | 2 weeks
  Before and after the intervention a mixed meal test will be performed
Changes in blood metabolome 1 week before, during 2 weeks of overfeeding and 2 weeks after overfeeding | 5 weeks
  Blood will be collected for metabolomics at screening, at baseline, during the overfeeding intervention and during the 2-week ad libitum intervention. Metabolomics will be performed using Mass Spectrometry.
Activity profile of 40 subjects during the 5 week study period | 5 weeks
  Assessment of daily physical activity levels (wearables and doubly-labelled water)
Detection of circulating factors | 5 weeks
  The investigators will measure the concentration of known circulating factors from fasted blood samples and from blood samples obtained during mixed meal test, such as: Glucose, insulin, hsCRP, Hba1c, cortisol, ACTH, lactate, fatty acids, triglycerides, glycerol, catecholamines, leptin, ghrelin, adiponectin, glucagon, GDF15, FGF21, FGF19, GIP, GLP-1, PYY, CCK, interleukins, cytokines, tissue-kines, T3, T4, TSH, cholesterol.
Gut microbiome profile before and after 14 days of overfeeding | 2 weeks
  Feces samples will be collected before and after 14 days of overfeeding and microbiome composition will be analyzed by using UPLC-MS/GC-MS.

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Clemmensen, Assoc. Prof., Principal Investigator — Assoc. prof. NNF Center for Basic Metabolic Research
Locations (1):
- University of Copenhagen, Copenhagen, Norrebro, Denmark